CLINICAL TRIAL: NCT03048201
Title: Post-market Registry Study on the Physica System Total Knee Replacement
Brief Title: Physica System Total Knee Replacement Registry Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-11
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee; Traumatic Arthritis; Avascular Necrosis; Degenerative Joint Disease of Knee; Rheumatoid Arthritis; Deformity of Knee
Keywords: Physica KR; Physica CR; Physica PS; Kinematic Retaining; Cruciate Retaining; Posterior Stabilized; Physica System
MeSH Terms: conditions — Osteoarthritis, Knee; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Subjects will receive a commercially available Physica system total knee replacement in one of 3 different configurations: KR (Kinematic Retaining), CR (Cruciate Retaining) and PS (Posterior Stabilized). The assignment of any patient involved in the study is determined by the aetiology preoperatively evaluated by the Investigator and falls within current practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Physica KR (Other): Subjects that receive the Physica Kinematic Retaining Knee System
  Interventions: Device: Physica Kinematic Retaining Knee System
- Physica CR (Other): Subjects that receive the Physica Cruciate Retaining Knee System
  Interventions: Device: Physica Cruciate Retaining Knee System
- Physica PS (Other): Subjects that receive the Physica Posterior Stabilized Knee System
  Interventions: Device: Physica Posterior Stabilized Knee System
- Physica CR with LMC Liner (Other): Subjects that receive the Physica Cruciate Retaining Knee System with LMC Liner
  Interventions: Device: Physica Cruciate Retaining Knee System with LMC Liner

INTERVENTIONS:
Device: Physica Kinematic Retaining Knee System — Modular total knee prosthesis with a Kinematic Retaining mechanism and posterior cruciate ligament (PCL) preservation
  Arms: Physica KR
Device: Physica Cruciate Retaining Knee System — Total knee prosthesis with posterior cruciate ligament (PCL) preservation
  Arms: Physica CR
Device: Physica Posterior Stabilized Knee System — Total knee prosthesis that sacrifices the posterior cruciate ligament (PCL) and replaces the functionality of the PCL with a post-cam mechanism.
  Arms: Physica PS
Device: Physica Cruciate Retaining Knee System with LMC Liner — Total knee prosthesis with posterior cruciate ligament (PCL) preservation
  Arms: Physica CR with LMC Liner

SUMMARY:
The primary objective of this study is to obtain long-term implant survivorship (out to 10 years) and to assess clinical, patient-reported outcome measures, and radiographic data for the commercially available Physica system. For ancillary arm, from baseline to 5-year follow-up.

DETAILED DESCRIPTION:
This is a post-market registry study; the study device is FDA cleared and used according to the intended use.

This is a multi-centre, prospective, non-randomized study.

Subjects will be implanted with one of the following configurations of the Physica system: Physica KR (Kinematic Retaining), Physica CR (Cruciate Retaining) or Physica PS (Posterior Stabilized). The assignment of any patient involved in the study is determined by the aetiology preoperatively evaluated by the Investigator and falls within current practice. The decision to use a specific prosthesis design is decided by the Investigators independently and clearly separated from the decision to include the patient in the study.

For the ancillary subgroup, investigators currently contributing to the primary patient group can also enroll additional patients to the ancillary subgroup. 3 existing sites and 2 additional sites are planned to be added to contribute to the additional 300 patients to be enrolled. These patients will follow the same study schedules as the main study, but follow-up is only up to 5 years.

Baseline measurements (pre-operative clinical analysis and radiographic analysis at 6-week FU) will serve as internal control term during the assessment of post-surgery data out to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of any race requiring a total knee replacement and suitable for the use of one of the configurations of the Physica system
2. Age> 22 (skeletally mature)
3. Patients who are suffering from non-inflammatory degenerative joint disease (NIDJD):

   including knee osteoarthritis, post-traumatic knee arthritis; or patients who are suffering from inflammatory arthritis; or patients that need correction of a functional deformity
4. Suitable candidates for TKR who have undamaged and functional collateral ligaments
5. Suitable candidates for TKR with Physica KR, CR, who have an undamaged and functional posterior cruciate ligament; or Physica LMC with or without a functioning posterior cruciate ligament or Physica PS with an absent or not-functioning posterior cruciate ligament and/or severe antero-posterior instability of the knee joint
6. Patients who understand the conditions of the study and are willing and able to comply with the prescribed rehabilitation and to perform all scheduled follow-up visits
7. Patients who have signed the Ethics Committee/IRB approved study-specific Informed Consent Form prior to the surgery

Exclusion Criteria:

1. Patients with severe instability of the knee joint secondary to the absence of collateral ligament integrity and/or function
2. Patients with active or any suspected infection (on the affected knee or systemic)
3. Previous partial knee replacement (unicompartimental, bicompartimental or patellofemoral joint replacement), patellectomy, high tibial osteotomy
4. Patients with significant bone loss on femoral or tibial joint side
5. Current treatment for malignant and/or life-threatening non-malignant disorders
6. Patients with known incompatibility or allergy to the product materials, and/or metal hypersensitivity to implant materials
7. Vascular insufficiency of lower limbs severe enough to interfere with the study evaluation
8. Patients with bone stock compromised by disease, infection or prior implantation that cannot provide adequate support and/or fixation to the prosthesis
9. Patients with systemic or metabolic disorders leading to progressive bone deterioration which may impair fixation and stability of the implant
10. Any concomitant disease and dependence that might affect the performance of the implanted prosthesis
11. Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation (e.g. primary osteoporosis with significant bone loss, haemophilic disease, septicaemia, persistent acute or chronic osteomyelitis)
12. Patients who have significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery and evaluation
13. Patients who have neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
14. Previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint
15. Any psychiatric illness that would prevent comprehension of the details and nature of the study
16. Patients currently participating in any other surgical intervention studies or pain management studies
17. Female patients who are pregnant, nursing, or planning a pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 10 years
  The primary endpoint is the definition of the implant survivorship of the study device to 10 years after the total knee replacement surgery.

SECONDARY OUTCOMES:
American Knee Society Score (KSS) 2011 | 10 years
  Clinical performance assessment measured by overall pain and functionality from baseline to 10-year follow-up
Patient-Reported Outcome Measures (PROMs) | 10 years
  Patient-Reported Outcome Measures (PROMs) including patient satisfaction achievement from baseline to 10-year follow-up
Radiographic Evaluation | 10 years
  • Radiographic implant evaluation and stability assessment from baseline to 10-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Pavan, Study Director — Limacorporate S.p.a
Locations (5):
- United States (5):
  - Eisenhower Desert Orthopedics Center - Harry and Diane Rinker Bldg, Rancho Mirage, California
  - The Orthopedics Clinic, Daytona Beach, Florida
  - Rush Castle Orthopaedics, Aurora, Illinois
  - Syracuse Orthopedic Specialists, Syracuse, New York
  - Joint Reconstructive Specialist, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No